CLINICAL TRIAL: NCT05375513
Title: A Home-based Personalized Multidomain RCT from the Canadian Therapeutic Platform for Multidomain Interventions to Prevent Dementia (CAN-THUMBS UP)
Brief Title: SYNERGIC-2 Trial (SYNchronizing, Exercises and Remedies to GaIn Cognition@home)
Acronym: SYN2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3948
Record Dates: First submitted 2022-04-21; First posted 2022-05-16 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-08

CONDITIONS: Mild Cognitive Impairment
Keywords: Dementia; Mild Cognitive Impairment; Virtual Interventions; Geriatric Medicine
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Intervention Model Description: The SYNERGIC-2 Trial is a single-blind, two-arm, randomized controlled trial (RCT) evaluating the cognitive effect of personalized multidomain interventions that target physical exercise, cognitive training, sleep, diet, and vascular risk factors. The SYNERGIC-2 Trial will be administered virtually through online video conferencing platform systems (WeBex or Zoom Healthcare©). Figure 1 illustrates the trial design. The trial adheres to the Consolidated Standards of Reporting Trials (CONSORT) guidelines for conducting and reporting clinical trials, as extended to non-pharmacological interventions. A total of 550 participants with MCI aged 60-85 will be enrolled and randomized into one of two arms, with 275 participants in each arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SYNERGIC 2 (Active Comparator): Personalized multidomain coached 1-to-1 interventions at home (PMI@Home) including:
  1. Physical Exercise
  2. Cognitive Training
  3. Diet
  4. Sleep
  5. Vascular Risk Factors Control
  Interventions: Other: PMI@Home
- Brain Health PRO (BHPro) (Placebo Comparator): Brain Health PRO (BHPROBHPRO) is an independent, educational program with content also related to:
  1. Physical Exercise
  2. Cognitive Training
  3. Diet
  4. Sleep
  5. Vascular Risk Factors
  6. Social engagement
  Interventions: Other: Brain Health Pro

INTERVENTIONS:
Other: PMI@Home — Personalized multidomain interventional program by combining tailored lifestyle interventions that targets 5 domains: physical activity, cognition, diet, sleep, and vascular risk factors. These interventions are tailored based on participants' baseline profile and progress in intensity following the principles of personalized medicine. All aspects of the PMI@home will be delivered remotely, at participants' homes, using a "digital platform" with scheduled bi-weekly 1-to1 coaching sessions. Delivery of interventions and assessments are centralized with 5 trained staff at the sponsor site (London) to assure logistics, standardization, and quality control.
  Arms: SYNERGIC 2
Other: Brain Health Pro — Online Modules:
  * Motivation, Self-Efficacy, Positive Health, Environment and Genetic risk
  * Physical Activity
  * Cognitively Stimulating Activities
  * Diet
  * Sleep
  * Social and Psychological Health
  * Vascular health
  * Vision and Hearing
  * Lifestyle Risk Impact Surveys
  * Goal Setting
  Arms: Brain Health PRO (BHPro)

SUMMARY:
In Canada, 1,700,000 adults are at risk of dementia, half of them with MCI,representing one of the largest groups at risk for an incurable disease. Epidemiological evidence suggests up to 40% of dementia cases might be preventable by targeting modifiable lifestyle and cardiovascular factors. Given that current treatments cannot modify the disease, prevention is critical. SYNERGIC-2 offers a "personalized multidomain intervention" that combines physical and cognitive training, sleep, diet, and vascular-metabolic interventions in individuals with MCI to synergistically enhance their overall brain health including cognition and contributes to maintaining their independence. Importantly, interventions will be provided at home using an existing virtual platform reducing delivery complexity and expanding the accessibility to a wider population, thus decreasing potential inequities. Improving older adults' brain health and achieving even a modest two-year dementia incidence delay will have a projected saving of $218 Billion in Canada's healthcare system over 30 years.

DETAILED DESCRIPTION:
Epidemiological evidence suggests up to 40% of potential dementia cases might be preventable by targeting modifiable lifestyle and cardiovascular factors; given that current treatments cannot modify the disease, prevention is a critical aspect. SYNERGIC-2 is the first large Canadian clinical trial using a 12-month home-based personalized multidomain lifestyle intervention to improve cognition in 550 older adults with Mild Cognitive Impairment (MCI), a pre-dementia state. These personalized at-home interventions target 5 domains with tailored physical exercise, cognitive training, diet recommendations, sleep interventions, and vascular risk factor management and are all delivered using a digital platform. Specifically, SYNERGIC-2 will be conducted with participants in their homes using video-conference meetings to test participants and to coach them 1-on-1 through the interventions on a web-based digital platform. The effect of these combined interventions on cognition will be compared to an online-educational program Brain Health PRO (BHPro). Both interventions are part of CAN-THUMBS UP, the interventional platform of the CCNA related to Canada Dementia Research Strategy; and constitutes Canada's contribution to the World-Wide-FINGERS Network. Importantly, these interventions have been selected because there is evidence that they synergistically enhance overall brain health including cognition and contributes to maintaining independence for individuals at risk for developing dementia.

ELIGIBILITY:
Inclusion Criteria

1. Ages 60-85 years.
2. Having mild cognitive impairment (MCI) defined as meeting all of the following:

   1. Presence of subjective memory complaints from the participant and/or informant.
   2. Objective impairment on cognitive tests independent of outcome measures.†
   3. Preserved activities of daily living assessed (>14/23 in Lawton-Brody IADL score). For the study, impairment of daily living will be assessed based on cognitive abilities, not physical abilities.
   4. Absence of clinical dementia per DSM-IV criteria †Objective cognitive impairment is operationalized as: Montreal Cognitive Assessment (MoCA) total score between 16 and 25 (inclusive), and/or RAVLT delayed recall ≤6, and /or Clinical Dementia Rating Scale (CDR) =0.5
3. Have ≥1 additional dementia risk factors targeted by our intervention as follows: low physical activity (less than 150 minutes of moderate-to-vigorous-intensity physical activity per week, as per GAQ), poor diet (14-item Mediterranean Diet Assessment (MDA-14) score ≤7), insomnia or subthreshold insomnia ( Insomnia Severity Index (ISI) score >7), and vascular-metabolic risk (Cardiovascular Risk Factors Aging and Incidence of Dementia (CAIDE) score ≥6 and/or diabetes (type I or II) and/or obesity (BMI≥30) and/or diagnosis of high blood pressure (hypertension) and/or smoking).
4. Have access to a home computer/laptop/tablet with home internet (have regular access to email) and ability to use technology (able to send and receive emails and join video conferences).
5. Self-reported levels of proficiency in English for speaking and understanding spoken and written language.
6. Have normal/corrected to normal vision in at least one eye to identify stimuli on computer/tablet screen.
7. Have normal to corrected hearing ability, in order for the participant to engage in digital/virtual communication. Research personnel will determine and assess the hearing ability as per participant's performance.
8. Able to comply with virtual visits, treatment plan, and trial-related activities.
9. Ability to participate in the study's exercise training as determined by the Get Active Questionnaire (GAQ).

Exclusion Criteria

1. Having a diagnosis of dementia (based on DSM-IV criteria).
2. Underlying severe disease that precludes engagement with interventions, including presence of psychiatric diagnoses (i.e., major depression (Geriatric Depression Scale (GDS-30) >19), schizophrenia, severe anxiety, neurological disorder with severe motor deficits, such as current parkinsonism or any neurological disorder with residual severe motor deficits (i.e., stroke with motor deficit), or presence of unstable (non-controlled e.g., symptoms that suggest instability or no treatment for their condition) chronic disease such as congestive heart failure (CHF), chronic obstructive pulmonary disease (COPD) that may preclude the participant from engaging properly with the trial interventions, or advanced-stage active cancer that at the study physician's discretion will prevent them from participating.
3. Having had surgery within the last 2 months or having an upcoming planned surgery in the next 12 months that could interfere with the participant's vision, hearing, mobility, or any other abilities to participate in the study.
4. Regular use of Benzodiazepine or neuroleptic drugs that may interfere with the participants ability to participate in the assessments and interventions.
5. Recent (in the past 12 months) and/or current substance or alcohol abuse.
6. Having had a transmural myocardial infarction (severe heart attack) within six months prior to enrollment in the clinical trial that according to the study physician may preclude physical activity performance.
7. Intention to enroll in other interventional clinical trials during same time.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in global cognition assessed using the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) with 13 items (ADASCog-13) | baseline and at 48 weeks (after interventions finalized)
  Global cognition will be assessed using the cognitive section of the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) with 13 items (ADASCog-13). This scale consists of 13 brief cognitive tests assessing attention, memory, language, executive function, praxis, orientation, and instrumental activities of daily living. The ADAS-Cog has been a significant outcome measure in numerous trials with MCI and AD to measure changes in cognitive performance in populations with cognitive impairment, it score ranges from 0 to 84, with higher scores indicating worse cognitive performance.

SECONDARY OUTCOMES:
Change in Anthropometric Measures | Baseline, month 3, mid-intervention at 6 months, month 9, and follow-up at 12 months
  Measurements of weight and hip/waist circumference will be done at home and self-reported by the participant. This can be used to characterize participant's body dimension and determine body mass index as kg/m^2 which can be used to estimate whether participants have obesity. A BMI greater than 30 is the cut off for obesity. Changes in waist circumference may also indicate visceral fat and cardiovascular risk.
Change in Cardiovascular Risk Factors, Aging, and Incidence of Dementia | Baseline, mid-intervention at 6 months, and follow-up at 12 months
  The Cardiovascular Risk Factors, Aging, and Incidence of Dementia (CAIDE) is a short questionnaire assessing midlife vascular risk for dementia, with scores ranging from 0 to 15 (higher scores suggesting higher risk) and has cut-off score of 5 for high risk.
Changes in the CCNA Gait Assessments results-Walking performance | Baseline, mid-intervention at 6 months, and follow-up at 12 months
  The CCNA gait assessment includes preferred and fast pace gait, and dual-task gait that comprises walking while performing three cognitively demanding tasks: counting backwards by ones, counting backwards by sevens, and naming animals. Participants will be asked to walk on a designated walking path(4 meters) in sight of camera
Changes in Clinical Dementia Rating scores | Baseline, mid-intervention at 6 months, and follow-up at 12 months
  The Clinical Dementia Rating (CDR) scale is a validated scale (0-3) used in longitudinal Alzheimer's Disease (AD) research to characterize the impact of cognitive decline on global function performance applicable to AD and related dementias. Information is obtained through a semi-structured interview of the patient and a reliable informant or collateral source (e.g. family member). A score of ) indicate no cognitive impairment; 0.5 for Mild cognitive impairment; 1 for early dementia; 2 for mild severe dementia; 3 for severe dementia
Changes in Digit Symbol Modalities Test - Oral Version (mental processing speed) | Baseline, mid-intervention at 6 months, and follow-up at 12 months
  The Digit Symbol Modalities Test is a 90-second, timed task that asks participants to orally match geometric figures with specific numbers according to a defined key (specifying which symbols are assigned to which numbers) that is provided at the top of the stimulus page. The oral Digit Symbol Modalities Test measures processing speed capabilities. The total number of numbers correctly matched with symbols is the final score for this test ranging from 0-110 correct numbers sequentially spoken.
Changes in Eating Pattern Self-Assessment | Baseline, month 3, mid-intervention at 6 months, month 9, and follow-up at 12 months
  The Eating Pattern Self-Assessment (EPSA) is a 12-item questionnaire assessing participants' dietary intake profiles over the past 12 months. No score provided
Changes in Fall Occurrence | Baseline, mid-intervention at 6 months, and follow-up at 12 months
  The monthly falls calendar that will be sent to help track any participant falls. Participants are being asked to complete this calendar on a daily basis in order to help investigators better track whether or not they have fallen since last intervention. A fall is defined as any unintentional event in which a participant falls to the ground or onto an object (e.g., a chair) no caused by a syncope or loss of consciousness. Total number of falls and consequences of falls is provided.
Changes in Generalized Anxiety Disorder (GAD-7) | Baseline, mid-intervention at 6 months, and follow-up at 12 months
  A questionnaire to score the frequency the participant experiences anxiety symptoms in the past 7 days with higher scores indicating worse anxiety symptoms. Score ranges from 0-21.
Change in Geriatric Depression Scale (GDS-30) | Baseline, mid-intervention at 6 months, and follow-up at 12 months
  A questionnaire to establish a participant's experience with depressive symptoms with higher score indicating more severe depressive symptoms. Score ranges from 0-30.
Change in Health Utility Index (HUI-3) | Baseline, mid-intervention at 6 months, and follow-up at 12 months
  The HUI-3 provides descriptive health profile measures on a generic scale with higher scores indicating better quality of life and global functionality. HUI also provides single-attribute scores of morbidities for the following attributes; vision, hearing, speech, ambulation, dexterity, emotion, cognition, and pain. Score ranges from one 1 to 6 or 1 to 5 depending on the domain; and sum of all domains could range from 8 to 45.
Changes in Health Resource Utilization Questionnaire (HRUQ) | Baseline, mid-intervention at 6 months, and follow-up at 12 months
  The HRUQ provides an overall assessment of a participants utilization of health-related resource use and costs for elderly adults with and without mild cognitive impairment.There is no scoring for the HRUQ
Changes in Insomnia Severity Index | Baseline, month 3, mid-intervention at 6 months, month 9, and follow-up at 12 months
  The Insomnia Severity Index (ISI) is a 7-item questionnaire assessing sleep onset, sleep maintenance, sleep satisfaction, and sleep problems.
Changes in International Physical Activity Questionnaire scores | Baseline, mid-intervention at 6 months, and follow-up at 12 months
  Modified for the elderly people, assesses older adults' level of physical activity, with a simple 7-item questionnaire. Scoring ranges from low, moderate and high.
Changes in the Lawton-Brody Instrumental Activities of Daily Living (IADL) scale | Baseline, mid-intervention at 6 months, and follow-up at 12 months
  Measures participant's ability to engage in instrumental activities of daily living via questionnaire assessing the ability to independently perform activities such as using the telephone, shopping, preparing meals, chores, household activities, managing prescriptions and medications, and managing personal finances. Score ranges from 0-23.
Changes in the Mediterranean Diet Assessment | Baseline, mid-intervention at 6 months, and follow-up at 12 months
  A 14-item questionnaire to help evaluate a participants Mediterranean ingredients in their diet. Score ranges from 0-14.
Changes in global cognitive function using Montreal Cognitive Assessment(MoCA) | Baseline, mid-intervention at 6 months, and follow-up at 12 months
  The MoCA is a brief screening instrument designed to detect global cognitive dysfunction. It assesses a range of different cognitive domains, including attention, executive functions, memory, language, visuo-constructional skills, abstract thinking, and orientation. Score ranges from 0-30.
Changes in the Oral Trail Making Test - Attention Shifting capabilities/executive functions using | Baseline, mid-intervention at 6 months, and follow-up at 12 months
  The Oral Trail Making Test (TMT) A & B is a two-part test that assesses attention speed, and mental flexibility and has been widely used in clinical settings for assessing deficits in attention and executive functioning. Score from part A ranges from 0-180; part B from 0-300 seconds. Longer times mean worse performance in the test.
Changes in Quality of Life Questionnaire (SF-36) | Baseline, mid-intervention at 6 months, and follow-up at 12 months
  The Short-Form Quality of Life Questionnaire (SF-36) is a 36-item questionnaire assessing quality of life, with scores ranging from 0 to 100 and higher scores indicating better quality of life.
Changes in Rey Auditory Verbal Learning Test (RAVLT)-Episodic memory | Baseline, mid-intervention at 6 months, and follow-up at 12 months
  The Rey Auditory Verbal Learning Test (RAVLT) assesses episodic memory, in which the participant is presented with 15 words in five presentations or trials, after which they are asked to recall the words (immediately and after a delay). Score ranges from 0 to 15 words recalled.
Changes in the Cognitive Expectancies Questionnaire | Baseline and follow-up at 12 months
  It is a version developed by the CCNA to measures participant's expectancies about the cognitive benefits of the intervention. Score ranges from 1 to 88. This questionnaire measures the participant's perception about the interventions. The questionnaire outcome is not related to participant's cognition, but participant's subjective perception about the interventions.
Changes in sleep pattern | Baseline, month 3, mid-intervention at 6 months, month 9, and follow-up at 12 months
  The Sleep Diary is self-administered of 10-days of sleep patterns to assess sleep quality and total of sleep time. It also helps to identify possible sleep disruptions that may affect sleep quality and identify certain habits that may explain sleeping issues.
Changes in physical activity in the elderly | Baseline, mid-intervention at 6 months, and follow-up at 12 months
  The Wrist (AX3) Accelerometer is used to detect movement, vibrations, and orientation changes to assess physical activity trends in older population.
Changes in behavior | Baseline, mid-intervention at 6 months, and follow-up at 12 months
  This questionnaire asks about eleven health behaviors, to be rated on a 0 (low) to 10 (high) scale. Prior research has demonstrated that a 1-point change on these 0 to 10 items is clinically meaningful.
Changes in BHPro questionnaires | Baseline, month 3, mid-intervention at 6 months, month 9, and follow-up at 12 months
  These questionnaires ask about cognition (6-item questionnaire), vascular health (4-item questionnaire), and social and psychological health (8-item questionnaire).
  * BHPro Questionnaire - Cognition: This questionnaire asks about participant's engagement in activities such as reading, crafting, and instrument playing. It does not provide any quantitative range score.
  * BHPro Questionnaire - Social and Psychological Health: This questionnaire asks about participant's emotions and mood. It does not provide any quantitative range score.
  * BHPro Questionnaire - Vascular Health: This questionnaire asks about participant's updated medical history. It does not provide any quantitative range score.
Changes in EEG | Baseline and follow-up at 12 months
  Participants will use the MUSE-S EEG Headband for 3 consecutive nights. The MUSE S Headband is a commercially available consumer headband that has 7 sensors, 2 on the forehead, 2 behind the ears, plus 3 reference sensors, to detect and measure EEG signals when sleeping.
Identification of APO-E variants, a planned panel of 31 single nucleotide polymorphisms (SNPs), and untargeted metabolomics | Baseline and follow-up at 12 months
  Participants will use the DNA-Genotek, which is a self-administered saliva collection kit to analyze saliva sample for possible identification of APO-E variants, a planned panel of 31 single nucleotide polymorphisms (SNPs), and untargeted metabolomics.
Changes in Resource Use Inventory Q7 & Q8 (RUI Q7 &Q8) | Baseline, mid-intervention at 6 months, and follow-up at 12 months
  Questions 7 and 8 from the Resource Use Inventory (RUI)28 questionnaire assess health-related resource use for caregivers. This instrument has been used for tracking resource use and costs in cognitively intact older adults, as well as with Alzheimer disease (AD). This is a self-report questionnaire investigates if participants received any help while preforming daily living tasks e.g., bathing, brushing, and getting the phone. It does not provide any quantitative range score.
Changes in 60s Chair Standing Test | Baseline, mid-intervention at 6 months, and follow-up at 12 months
  Participants will be performing the one-minute chair stand test while being assessed via video conferencing by a research team member to evaluate mobility.
Changes in The Activities-specific Balance Confidence Scale (ABC) questionnaire | Baseline, mid-intervention at 6 months, and follow-up at 12 months
  The ABC questionnaire consists of 16 questions where the participants rate their confidence that they will not lose their balance or become unsteady while performing different activities. They need to rate 16 different activities from 0 to 100, 0 being not confident at all, and 100 being completely confident on their abilities to perform the activity.
Changes in The Short Physical Performance Battery (SPPB) | Baseline, mid-intervention at 6 months, and follow-up at 12 months
  The SPPB is an objective assessment tool for evaluating lower extremity functioning in older adults. Score ranges from 0 to 12. 0 being frail (disabled), and 12 being no mobility disability issues.

OTHER OUTCOMES:
Recruitment Rate | Throughout study completion - avg. 12 months/participant
  Defined as the total percent of enrolled participants relative to the number of people screened for eligibility. Score is calculated as the ratio of screened and enrolled participants per month. Higher scores = better recruitment rates.
Retention Rate | Throughout study completion - avg. 12 months/participant
  Defined as the total percent of enrolled participants who continue throughout the trial and participate in outcomes assessments as follows:
  * Enrollment retention: of those enrolled participants, the % who complete immediate 6-month post intervention assessment, and;
  * Follow-up retention: of those who complete the immediate 6-month post intervention follow-up assessment, the % of participants who complete the 6-month post-intervention follow-up assessment at 12-months.
Assessment Tolerability | Baseline
  Defined as total percent of participants not voluntarily dropping out during baseline or between baseline assessment and prior to allocation to intervention group.
Adverse Events | Throughout study completion - avg. 12 months/participant
  Frequency cross-tabulation of AE severity versus AE relation to trial
Data Loss | Throughout study completion - avg. 12 months/participant
  Defined as data lost due to technical failures, personnel errors or participant non-compliance and is calculated as percentages.
Sex of Participant | Baseline
  This measurement will be self-reported.
Age of Participant | Baseline
  This measurement will be self-reported.
Medications Taken by Participant | Baseline, mid-intervention at 6 months, and follow-up at 12 months
  This measurement will be self-reported. And will be reported as individuals medications and total amount.
Chronic Diseases of Participant | Baseline, mid-intervention at 6 months, and follow-up at 12 months
  This measurement will be self-reported and will be monitored throughout the trial

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Montero-Odasso, MD, PhD, Principal Investigator — St. Joseph's Health Care London, Parkwood Hospital
Locations (8):
- Canada (8):
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - University of New Brunswick, Fredericton, New Brunswick
  - St. Joseph's Health Care London, Parkwood Hospital, London, Ontario
  - University of Ottawa, Ottawa, Ontario
  - Baycrest Academy for Research and Education, Toronto, Ontario
  - University of Waterloo, Waterloo, Ontario
  - Concordia University, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Delis DC, Kramer JH, Kaplan E, Holdnack J. Reliability and validity of the Delis-Kaplan Executive Function System: an update. J Int Neuropsychol Soc. 2004 Mar;10(2):301-3. doi: 10.1017/S1355617704102191. No abstract available. PMID 15012851
- [Background] Schmidt M. Rey auditory verbal learning test: A handbook. Los Angeles, CA: Western Psychological Services.; 1996.
- [Background] Esther Strauss OS. Trail Making Tests. New York: Oxford University Press; 1998.
- [Background] Koblinsky ND, Anderson ND, Ajwani F, Parrott MD, Dawson D, Marzolini S, Oh P, MacIntosh B, Middleton L, Ferland G, Greenwood CE. Feasibility and preliminary efficacy of the LEAD trial: a cluster randomized controlled lifestyle intervention to improve hippocampal volume in older adults at-risk for dementia. Pilot Feasibility Stud. 2022 Feb 9;8(1):37. doi: 10.1186/s40814-022-00977-6. PMID 35139918
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] DOPPELT JE, WALLACE WL. Standardization of the Wechsler adult intelligence scale for older persons. J Abnorm Psychol. 1955 Sep;51(2):312-30. doi: 10.1037/h0044391. No abstract available. PMID 13263050
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Peters R, Booth A, Rockwood K, Peters J, D'Este C, Anstey KJ. Combining modifiable risk factors and risk of dementia: a systematic review and meta-analysis. BMJ Open. 2019 Jan 25;9(1):e022846. doi: 10.1136/bmjopen-2018-022846. PMID 30782689
- [Background] Bennett DA, Schneider JA, Buchman AS, Barnes LL, Boyle PA, Wilson RS. Overview and findings from the rush Memory and Aging Project. Curr Alzheimer Res. 2012 Jul;9(6):646-63. doi: 10.2174/156720512801322663. PMID 22471867
- [Background] Falck RS, Davis JC, Best JR, Li LC, Chan PCY, Wyrough AB, Landry GJ, Liu-Ambrose T. Buying time: a proof-of-concept randomized controlled trial to improve sleep quality and cognitive function among older adults with mild cognitive impairment. Trials. 2018 Aug 17;19(1):445. doi: 10.1186/s13063-018-2837-7. PMID 30119694
- [Background] Carney CE, Buysse DJ, Ancoli-Israel S, Edinger JD, Krystal AD, Lichstein KL, Morin CM. The consensus sleep diary: standardizing prospective sleep self-monitoring. Sleep. 2012 Feb 1;35(2):287-302. doi: 10.5665/sleep.1642. PMID 22294820
- [Background] Csizmadi I, Kahle L, Ullman R, Dawe U, Zimmerman TP, Friedenreich CM, Bryant H, Subar AF. Adaptation and evaluation of the National Cancer Institute's Diet History Questionnaire and nutrient database for Canadian populations. Public Health Nutr. 2007 Jan;10(1):88-96. doi: 10.1017/S1368980007184287. PMID 17212847
- [Background] Sala-Vila A, Valls-Pedret C, Rajaram S, Coll-Padros N, Cofan M, Serra-Mir M, Perez-Heras AM, Roth I, Freitas-Simoes TM, Domenech M, Calvo C, Lopez-Illamola A, Bitok E, Buxton NK, Huey L, Arechiga A, Oda K, Lee GJ, Corella D, Vaque-Alcazar L, Sala-Llonch R, Bartres-Faz D, Sabate J, Ros E. Effect of a 2-year diet intervention with walnuts on cognitive decline. The Walnuts And Healthy Aging (WAHA) study: a randomized controlled trial. Am J Clin Nutr. 2020 Mar 1;111(3):590-600. doi: 10.1093/ajcn/nqz328. PMID 31912155
- [Background] Loughrey DG, Lavecchia S, Brennan S, Lawlor BA, Kelly ME. The Impact of the Mediterranean Diet on the Cognitive Functioning of Healthy Older Adults: A Systematic Review and Meta-Analysis. Adv Nutr. 2017 Jul 14;8(4):571-586. doi: 10.3945/an.117.015495. Print 2017 Jul. PMID 28710144
- [Background] Borm GF, Fransen J, Lemmens WA. A simple sample size formula for analysis of covariance in randomized clinical trials. J Clin Epidemiol. 2007 Dec;60(12):1234-8. doi: 10.1016/j.jclinepi.2007.02.006. Epub 2007 Jun 6. PMID 17998077
- [Background] Petrella AFM, Gill DP, Petrella RJ. Evaluation of the Get Active Questionnaire in community-dwelling older adults. Appl Physiol Nutr Metab. 2018 Jun;43(6):587-594. doi: 10.1139/apnm-2017-0489. Epub 2018 Jan 17. PMID 29342366
- [Background] Cassarly C, Matthews LJ, Simpson AN, Dubno JR. The Revised Hearing Handicap Inventory and Screening Tool Based on Psychometric Reevaluation of the Hearing Handicap Inventories for the Elderly and Adults. Ear Hear. 2020 Jan/Feb;41(1):95-105. doi: 10.1097/AUD.0000000000000746. PMID 31124792
- [Background] Stephen R, Liu Y, Ngandu T, Rinne JO, Kemppainen N, Parkkola R, Laatikainen T, Paajanen T, Hanninen T, Strandberg T, Antikainen R, Tuomilehto J, Keinanen Kiukaanniemi S, Vanninen R, Helisalmi S, Levalahti E, Kivipelto M, Soininen H, Solomon A. Associations of CAIDE Dementia Risk Score with MRI, PIB-PET measures, and cognition. J Alzheimers Dis. 2017;59(2):695-705. doi: 10.3233/JAD-170092. PMID 28671114
- [Background] Sindi S, Calov E, Fokkens J, Ngandu T, Soininen H, Tuomilehto J, Kivipelto M. The CAIDE Dementia Risk Score App: The development of an evidence-based mobile application to predict the risk of dementia. Alzheimers Dement (Amst). 2015 Jul 2;1(3):328-33. doi: 10.1016/j.dadm.2015.06.005. eCollection 2015 Sep. PMID 27239514
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Martinez-Gonzalez MA, Garcia-Arellano A, Toledo E, Salas-Salvado J, Buil-Cosiales P, Corella D, Covas MI, Schroder H, Aros F, Gomez-Gracia E, Fiol M, Ruiz-Gutierrez V, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Munoz MA, Warnberg J, Ros E, Estruch R; PREDIMED Study Investigators. A 14-item Mediterranean diet assessment tool and obesity indexes among high-risk subjects: the PREDIMED trial. PLoS One. 2012;7(8):e43134. doi: 10.1371/journal.pone.0043134. Epub 2012 Aug 14. PMID 22905215
- [Background] Feeny D, Furlong W, Torrance GW, Goldsmith CH, Zhu Z, DePauw S, Denton M, Boyle M. Multiattribute and single-attribute utility functions for the health utilities index mark 3 system. Med Care. 2002 Feb;40(2):113-28. doi: 10.1097/00005650-200202000-00006. PMID 11802084
- [Background] Lyons RA, Perry HM, Littlepage BN. Evidence for the validity of the Short-form 36 Questionnaire (SF-36) in an elderly population. Age Ageing. 1994 May;23(3):182-4. doi: 10.1093/ageing/23.3.182. PMID 8085500
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Background] Morris JC. The Clinical Dementia Rating (CDR): current version and scoring rules. Neurology. 1993 Nov;43(11):2412-4. doi: 10.1212/wnl.43.11.2412-a. No abstract available. PMID 8232972
- [Background] Dawidowicz L, L Ash E, Korczyn AD, Andelman F, Levy S, Elkana O. Can the RAVLT predict deterioration from MCI to dementia? Data from long term follow up. Exp Aging Res. 2021 Jul-Sep;47(4):347-356. doi: 10.1080/0361073X.2021.1898182. Epub 2021 Mar 11. PMID 33704020
- [Background] Berrigan LI, Fisk JD, Walker LA, Wojtowicz M, Rees LM, Freedman MS, Marrie RA. Reliability of regression-based normative data for the oral symbol digit modalities test: an evaluation of demographic influences, construct validity, and impairment classification rates in multiple sclerosis samples. Clin Neuropsychol. 2014;28(2):281-99. doi: 10.1080/13854046.2013.871337. Epub 2014 Jan 20. PMID 24438521
- [Background] Ricker JH, Axelrod BN. Analysis of an Oral Paradigm for the Trail Making Test. Assessment. 1994 Mar;1(1):47-52. doi: 10.1177/1073191194001001007. PMID 9463499
- [Background] Chapman JE, Cadilhac DA, Gardner B, Ponsford J, Bhalla R, Stolwyk RJ. Comparing face-to-face and videoconference completion of the Montreal Cognitive Assessment (MoCA) in community-based survivors of stroke. J Telemed Telecare. 2021 Sep;27(8):484-492. doi: 10.1177/1357633X19890788. Epub 2019 Dec 9. PMID 31813317
- [Background] Takeda A, Loveman E, Clegg A, Kirby J, Picot J, Payne E, Green C. A systematic review of the clinical effectiveness of donepezil, rivastigmine and galantamine on cognition, quality of life and adverse events in Alzheimer's disease. Int J Geriatr Psychiatry. 2006 Jan;21(1):17-28. doi: 10.1002/gps.1402. PMID 16323253
- [Background] Yoshida K, Yamaoka Y, Eguchi Y, Sato D, Iiboshi K, Kishimoto M, Mimura M, Kishimoto T. Remote neuropsychological assessment of elderly Japanese population using the Alzheimer's Disease Assessment Scale: A validation study. J Telemed Telecare. 2020 Aug-Sep;26(7-8):482-487. doi: 10.1177/1357633X19845278. Epub 2019 May 8. PMID 31068063
- [Background] Montero-Odasso M, Almeida QJ, Burhan AM, Camicioli R, Doyon J, Fraser S, Li K, Liu-Ambrose T, Middleton L, Muir-Hunter S, McIlroy W, Morais JA, Pieruccini-Faria F, Shoemaker K, Speechley M, Vasudev A, Zou GY, Berryman N, Lussier M, Vanderhaeghe L, Bherer L. SYNERGIC TRIAL (SYNchronizing Exercises, Remedies in Gait and Cognition) a multi-Centre randomized controlled double blind trial to improve gait and cognition in mild cognitive impairment. BMC Geriatr. 2018 Apr 16;18(1):93. doi: 10.1186/s12877-018-0782-7. PMID 29661156
- [Background] Kueper JK, Speechley M, Montero-Odasso M. The Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog): Modifications and Responsiveness in Pre-Dementia Populations. A Narrative Review. J Alzheimers Dis. 2018;63(2):423-444. doi: 10.3233/JAD-170991. PMID 29660938
- [Background] Norton S, Matthews FE, Barnes DE, Yaffe K, Brayne C. Potential for primary prevention of Alzheimer's disease: an analysis of population-based data. Lancet Neurol. 2014 Aug;13(8):788-94. doi: 10.1016/S1474-4422(14)70136-X. PMID 25030513
- [Background] Solomon A, Mangialasche F, Richard E, Andrieu S, Bennett DA, Breteler M, Fratiglioni L, Hooshmand B, Khachaturian AS, Schneider LS, Skoog I, Kivipelto M. Advances in the prevention of Alzheimer's disease and dementia. J Intern Med. 2014 Mar;275(3):229-50. doi: 10.1111/joim.12178. PMID 24605807
- [Background] Richards M, Deary IJ. A life course approach to cognitive reserve: a model for cognitive aging and development? Ann Neurol. 2005 Oct;58(4):617-22. doi: 10.1002/ana.20637. PMID 16178025
- [Background] Ngandu T, Lehtisalo J, Solomon A, Levalahti E, Ahtiluoto S, Antikainen R, Backman L, Hanninen T, Jula A, Laatikainen T, Lindstrom J, Mangialasche F, Paajanen T, Pajala S, Peltonen M, Rauramaa R, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Soininen H, Kivipelto M. A 2 year multidomain intervention of diet, exercise, cognitive training, and vascular risk monitoring versus control to prevent cognitive decline in at-risk elderly people (FINGER): a randomised controlled trial. Lancet. 2015 Jun 6;385(9984):2255-63. doi: 10.1016/S0140-6736(15)60461-5. Epub 2015 Mar 12. PMID 25771249
- [Background] Orgeta V, Mukadam N, Sommerlad A, Livingston G. The Lancet Commission on Dementia Prevention, Intervention, and Care: a call for action. Ir J Psychol Med. 2019 Jun;36(2):85-88. doi: 10.1017/ipm.2018.4. PMID 31187723
- [Background] Anstey KJ, Peters R, Zheng L, Barnes DE, Brayne C, Brodaty H, Chalmers J, Clare L, Dixon RA, Dodge H, Lautenschlager NT, Middleton LE, Qiu C, Rees G, Shahar S, Yaffe K. Future Directions for Dementia Risk Reduction and Prevention Research: An International Research Network on Dementia Prevention Consensus. J Alzheimers Dis. 2020;78(1):3-12. doi: 10.3233/JAD-200674. PMID 32925063
- [Background] Wilson RS, Leurgans SE, Boyle PA, Schneider JA, Bennett DA. Neurodegenerative basis of age-related cognitive decline. Neurology. 2010 Sep 21;75(12):1070-8. doi: 10.1212/WNL.0b013e3181f39adc. Epub 2010 Sep 15. PMID 20844243
- [Background] James BD, Bennett DA. Causes and Patterns of Dementia: An Update in the Era of Redefining Alzheimer's Disease. Annu Rev Public Health. 2019 Apr 1;40:65-84. doi: 10.1146/annurev-publhealth-040218-043758. Epub 2019 Jan 14. PMID 30642228
- [Background] Diagnostic And Statistical Manual of Mental Disorders : DSM-IV. Washington DC: American Psychiatric Association; 1994.
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Albert MS, DeKosky ST, Dickson D, Dubois B, Feldman HH, Fox NC, Gamst A, Holtzman DM, Jagust WJ, Petersen RC, Snyder PJ, Carrillo MC, Thies B, Phelps CH. The diagnosis of mild cognitive impairment due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):270-9. doi: 10.1016/j.jalz.2011.03.008. Epub 2011 Apr 21. PMID 21514249
- [Background] Rising the Tide: The Impact of Dementia on Canadian Society. 2012.
- [Background] Kivipelto M, Mangialasche F, Snyder HM, Allegri R, Andrieu S, Arai H, Baker L, Belleville S, Brodaty H, Brucki SM, Calandri I, Caramelli P, Chen C, Chertkow H, Chew E, Choi SH, Chowdhary N, Crivelli L, Torre R, Du Y, Dua T, Espeland M, Feldman HH, Hartmanis M, Hartmann T, Heffernan M, Henry CJ, Hong CH, Hakansson K, Iwatsubo T, Jeong JH, Jimenez-Maggiora G, Koo EH, Launer LJ, Lehtisalo J, Lopera F, Martinez-Lage P, Martins R, Middleton L, Molinuevo JL, Montero-Odasso M, Moon SY, Morales-Perez K, Nitrini R, Nygaard HB, Park YK, Peltonen M, Qiu C, Quiroz YT, Raman R, Rao N, Ravindranath V, Rosenberg A, Sakurai T, Salinas RM, Scheltens P, Sevlever G, Soininen H, Sosa AL, Suemoto CK, Tainta-Cuezva M, Velilla L, Wang Y, Whitmer R, Xu X, Bain LJ, Solomon A, Ngandu T, Carrillo MC. World-Wide FINGERS Network: A global approach to risk reduction and prevention of dementia. Alzheimers Dement. 2020 Jul;16(7):1078-1094. doi: 10.1002/alz.12123. Epub 2020 Jul 5. PMID 32627328
- [Background] Montero-Odasso M, Ismail Z, Livingston G. One third of dementia cases can be prevented within the next 25 years by tackling risk factors. The case "for" and "against". Alzheimers Res Ther. 2020 Jul 8;12(1):81. doi: 10.1186/s13195-020-00646-x. PMID 32641088
- [Background] Livingston G, Huntley J, Sommerlad A, Ames D, Ballard C, Banerjee S, Brayne C, Burns A, Cohen-Mansfield J, Cooper C, Costafreda SG, Dias A, Fox N, Gitlin LN, Howard R, Kales HC, Kivimaki M, Larson EB, Ogunniyi A, Orgeta V, Ritchie K, Rockwood K, Sampson EL, Samus Q, Schneider LS, Selbaek G, Teri L, Mukadam N. Dementia prevention, intervention, and care: 2020 report of the Lancet Commission. Lancet. 2020 Aug 8;396(10248):413-446. doi: 10.1016/S0140-6736(20)30367-6. Epub 2020 Jul 30. No abstract available. PMID 32738937
- [Background] Alzheimer Society of Canada. Report summary Prevalence and monetary costs of dementia in Canada (2016): a report by the Alzheimer Society of Canada. Health Promot Chronic Dis Prev Can. 2016 Oct;36(10):231-232. PMID 27768560